CLINICAL TRIAL: NCT00037869
Title: High Dose I-131 Metaiodobenzylguanidine (MIBG) Therapy for Metastatic Neuroendocrine Tumors
Brief Title: High Dose I-131 Metaiodobenzylguanidine(MIBG) for Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-063
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Neuroendocrine Tumors; Metastases, Neoplasm
Keywords: Metastatic neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasm Metastasis | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIBG (Experimental): High Dose I-131 Metaiodobenzylguanidine
  Interventions: Drug: I-131 Metaiodobenzylguanidine

INTERVENTIONS:
Drug: I-131 Metaiodobenzylguanidine
  Other Names: MIBG

SUMMARY:
The goal of this clinical research study is to learn if I-131 Metaiodobenzylguanidine (MIBG) can shrink or slow the growth of the tumor(s) in patients with metastatic neuroendocrine tumors. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
MIBG is used to visualize a group of specific cells in the body. It has been known to deliver the radioactive iodine to the tumor (cancer) cells selectively and result in their destruction.

Before treatment starts, patients will be evaluated with a tracer scan, using either I-131 MIBG or I-123 MIBG to locate the tumor site(s). If no MIBG accumulation can be found within tumor sites, the patient will not be able to continue on this study. Patients will also have CT scans and urine and blood tests. Women able to have children will have a pregnancy test.

If tumor sites are found and patients are fully eligible, they will receive a therapeutic (treatment) dose of I-131 MIBG by vein over 120 minutes. Some patients may have to receive a lower dose of MIBG. Patients will require hospitalization for treatment and will remain hospitalized for about 3-6 days.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 years of age and older
* Sex: male or female; female patients with child bearing potential must have a negative serum HCG pregnancy test within 72 hours prior to treatment;
* Diagnostic criteria- Patients must meet all of the following:

  1. Histologically documented neuroendocrine tumor.
  2. Labeled MIBG concentration in the tumor site(s) on diagnostic scan.
  3. good to excellent performance status.
* A patient for whom written voluntary informed consent has been obtained prior to study and participation.
* Patients can have had prior chemotherapy, as long as hematological parameters meet specifications.
* Please refer to Appendix D Drugs and Other Interactions for list of medications patient needs to cease 2 weeks prior to therapy. Patient should check with primary physician after therapy about resuming these medications.
* Patients with treatment refractory or relapsed advanced or disease not amendable to significant response (>25% to available chemotherapy) or metastatic disease not amenable to standard therapy.

Exclusion Criteria:

* Patients with inadequate hematopoietic bone marrow function: ANC<1000 cells/mm3, or platelets<75k cells/mm3 or hemoglobin<10g/dL.
* Patients with impaired renal function: creatinine>1.5mg/dL.
* Patients with impaired hepatic function: AST or ALT > 3.0 X upper limit of normal or total bilirubin > 2.0 mg/dL.
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at time of study entry.
* Female patients who are breast-feeding.
* Children less than 2 years of age.
* Patients with previous total body irradiation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2001-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Podoloff, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States